CLINICAL TRIAL: NCT04424069
Title: Optical Coherence Tomography Angiography Analysis of Macular and Papillary Perfusion After Variable Refractive Surgery Methods in Myopic Patients
Brief Title: OCTA Analysis of Macular and Papillary Perfusion After Refractive Surgery in Myopes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Abdelfattah Sorour, Retina consultant & the principal investigator, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 33553/12/19
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Myopia; Perfusion; Complications
MeSH Terms: conditions — Myopia | interventions — Refractive Surgical Procedures

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LASIK group (Active Comparator): Patients will do excimer laser LASIK operation for correction of myopia with flap creation by mechanical keratome
  Interventions: Procedure: Refractive surgery
- SMILE group (Active Comparator): Patients will do Femtosecond laser assisted corneal refractive surgery for correction of myopia
  Interventions: Procedure: Refractive surgery
- Photorefractive keratectomy group (Active Comparator): Patients that will undergo photorefractive keratectomy for correction of myopia
  Interventions: Procedure: Refractive surgery
- Refractive lens exchange (Active Comparator): Include eyes that will undergo refractive lens exchange
  Interventions: Procedure: Refractive surgery
- Control group (No Intervention): Myopic control eyes with no surgical intervention

INTERVENTIONS:
Procedure: Refractive surgery — Myopic patients seeking refractive surgery will be assigned to the study groups to assess the change in myopic and papillary perfusion in these different prodecures
  Arms: LASIK group; Photorefractive keratectomy group; Refractive lens exchange; SMILE group

SUMMARY:
Refractive surgery for correction of myopia is very common nowadays. However, various refractive techniques may be associated with increase in the IOP, especially during flap creation. It is assumed that marked intraoperative IOP increase lead to macular and optic disc head circulation compromise. The purpose of this study is to assess the change of macular and papillary perfusion, using optical coherence tomography angiography (OCTA) imaging of the macula and optic disc of myopic patients before and after various refractive surgery methods.

DETAILED DESCRIPTION:
Myopia is the most prevalent ocular disorder in children worldwide, and one of the major causes of visual deterioration in all age groups. Highest prevalence rates are in East Asian countries (affecting up to 83% of Singaporean teenagers), however, it is very common in all other countries. While mild to moderate myopia usually stabilizes within the third decade, pathological myopia is associated with progressive globe elongation, and development of various macular complications including; foveoschisis, choroidal neovascularization (CNV), myopic macular hole, and myopic vitreomacular traction (VMT).

Refractive surgery has become popular for correcting ametropia including myopia. Most commonly used refractive procedures include corneal refractive surgeries especially laser in-situ keratomileusis (LASIK), and Photorefractive keratectomy (PRK), Phakic Intraocular Lenses (Phakic IOLs) and refractive lens exchange.

In LASIK, the creation of a corneal lamellar flap requires placement of a suction ring on the anterior segment of the eye, which transiently elevates the intraocular pressure (IOP) to levels exceeding 65 mmHg. Experimental studies in animal eyes have found that the IOP can increase to between 80 mmHg and 360 mmHg during this vacuum phase and lamellar cut with the microkeratome. Recent advances utilizing the femtosecond laser may serve as an alternative to the mechanical microkeratome, with a low-pressure suction ring. In studies using porcine eyes, the IOP during the suctioning or laser application phase reached a maximum of 135 mmHg using the femtosecond laser, lower than pressures reached with a traditional microkeratome, but for a longer duration of time. Similarly in refractive lens procedures, intraoperative IOP was found to exceed 60 mmHg.

Intraocular pressure elevation during refractive procedures may cause a reduction in the perfusion of the retina and optic nerve head, posterior displacement of the lamina cribrosa, and a decline in ocular perfusion pressure of the posterior ciliary arteries. Although this IOP elevation is temporary, the potential for ischemic or pressure-induced damage to the optic nerve head and the retinal nerve fiber layer exists.

Optical coherence tomography angiography (OCTA) is a recent noninvasive imaging technique that allows for volumetric visualization of eye vasculature. OCTA has shown promise in better elucidating the pathophysiology of several retinal vascular diseases. Swept-source OCTA uses long wavelength ̰ 1,050nm, which can penetrate through deeper layers of the eye and can traverse opacities of media such as cataracts, hemorrhages and vitreous opacities [6]. Optical coherence tomographic angiograms can further be manually or automatically segmented with preprogrammed software to highlight individual layers of the retina, optic nerve head choriocapillaris, and choroid. The user can either analyze en face images extending from the inner limiting membrane to choroid or use automated views to locate a vascular or structural lesion within the retina.

The purpose of this study is to assess the change of macular and papillary perfusion, using optical coherence tomography angiography (OCTA) imaging of the macula and optic disc of myopic patients subject to various refractive surgery methods. We will compare between these methods to evaluate which one is associated with least adverse effect on ocular perfusion. To date no such evaluation has been done using OCTA, because of relatively recent onset of this technology. Traditional imaging methods such as color fundus photography and fluorescein angiography have limited resolution for retinal vasculature that mad such evaluation in the past using these methods not feasible, however, OCTA is very promising for the proper analysis of changes in the ocular perfusion. Results of this study will have significant clinical and practical implications and may change the approach for surgical correction of such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 20 - 35 years
2. Patients: who are seeking and fit for refractive surgery
3. Spherical equivalent refractive error: between (-2 to -9 D)

Exclusion Criteria:

1. Maculopathies (hereditary or acquired)
2. optic nerve head pathologies (tilted disc, drusen, optic disc edema, atrophy, etc.)
3. optic neuropathies (demyelinating, infectious, ischemic, etc.)
4. adjusted IOP for central corneal thickness more than 21 mmHg
5. surgery-induced corneal edema
6. dense cataracts that can disrupt images
7. systemic diseases (vasculitis, diabetes mellitus, hypertension, etc.)
8. any previous ocular surgery,
9. patients with bad quality images or complicated surgeries will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Vessel density from enface OCT angiogram | 6 months
  VD analysis computes the percentage of area occupied by OCTA detected vasculature in a measured area

CONTACTS AND LOCATIONS:
Overall Officials: Rauf A gaber, MD, Study Chair — Tanta University
Locations (1):
- Ophthalmology Department, Faculty of medicine, Tanta Univeristy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flitcroft DI, He M, Jonas JB, Jong M, Naidoo K, Ohno-Matsui K, Rahi J, Resnikoff S, Vitale S, Yannuzzi L. IMI - Defining and Classifying Myopia: A Proposed Set of Standards for Clinical and Epidemiologic Studies. Invest Ophthalmol Vis Sci. 2019 Feb 28;60(3):M20-M30. doi: 10.1167/iovs.18-25957. PMID 30817826
- [Background] Renones de Abajo J, Estevez Jorge B, Gonzalez Martin JM, Carreras Diaz H, Loro Ferrer JF, Anton Lopez A. Effect of femtosecond laser-assisted lens surgery on the optic nerve head and the macula. Int J Ophthalmol. 2019 Jun 18;12(6):961-966. doi: 10.18240/ijo.2019.06.13. eCollection 2019. PMID 31236353
- [Background] Vetter JM, Schirra A, Garcia-Bardon D, Lorenz K, Weingartner WE, Sekundo W. Comparison of intraocular pressure during corneal flap preparation between a femtosecond laser and a mechanical microkeratome in porcine eyes. Cornea. 2011 Oct;30(10):1150-4. doi: 10.1097/ICO.0b013e318212110a. PMID 21912236
- [Background] Khng C, Packer M, Fine IH, Hoffman RS, Moreira FB. Intraocular pressure during phacoemulsification. J Cataract Refract Surg. 2006 Feb;32(2):301-8. doi: 10.1016/j.jcrs.2005.08.062. PMID 16565009
- [Background] Whitson JT, McCulley JP, Cavanagh HD, Song J, Bowman RW, Hertzog L. Effect of laser in situ keratomileusis on optic nerve head topography and retinal nerve fiber layer thickness. J Cataract Refract Surg. 2003 Dec;29(12):2302-5. doi: 10.1016/s0886-3350(03)00466-8. PMID 14709290
- [Background] Or C, Sabrosa AS, Sorour O, Arya M, Waheed N. Use of OCTA, FA, and Ultra-Widefield Imaging in Quantifying Retinal Ischemia: A Review. Asia Pac J Ophthalmol (Phila). 2018 Jan-Feb;7(1):46-51. doi: 10.22608/APO.201812. Epub 2018 Feb 13. PMID 29436208